CLINICAL TRIAL: NCT06752915
Title: The Aim of This Study is to Determine the Effect of Acupressure Applied to Individuals with COPD on Dyspnea and Anxiety: It is Important for the Transfer of Nonpharmacological Methods to Clinical Applications
Brief Title: The Effect of Acupressure on Dyspnea and Anxiety Levels
Acronym: nursing
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ÇİĞDEM ERGİN (Other)
Responsible Party: Sponsor-Investigator, ÇİĞDEM ERGİN, PhD student and nursing, Cukurova University
Organization: Cukurova University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 0000-0002-3458-1670
Record Dates: First submitted 2024-12-09; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Simple randomization was used in the study. By computer randomization, patients were divided into intervention and control groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- acupressure (Experimental): The intervention group will receive acupressure at points LI4, HT7, LU1 and ST36, two minutes, once a day, 5 days a week, for 1 month.
  Interventions: Behavioral: acupressure application
- control group (No Intervention): No application will be made to the control group. Only pre-test and post-test will be applied.

INTERVENTIONS:
Behavioral: acupressure application — Acupressure massage will be applied to LI4, HT7, LU1 and ST 36 acupuncture points for 2 minutes.
  Arms: acupressure

SUMMARY:
The aim of this study is to determine the effect of acupressure applied to individuals with COPD on dyspnea and anxiety. It is important for the transfer of nonpharmacological methods to clinical applications.

DETAILED DESCRIPTION:
The pathophysiological changes that occur in the airways and alveoli in chronic obstructive pulmonary disease can cause many symptoms such as dyspnea, cough and sputum, which restrict the daily lives of individuals. Dyspnea and anxiety are at the top of the list among these symptoms, which affect individuals in many ways and limit them in many areas. While physiological, psychological and sociological factors cause dyspnea, the anxiety that develops in patients along with dyspnea also accompanies the symptoms. These symptoms seen in individuals with COPD not only negatively affect the quality of life of individuals, but also bring about psychological, cognitive, economic and social problems. Therefore, reducing anxiety and dyspnea in patients with COPD is of great importance in controlling the symptoms. Recently, acupressure has been frequently preferred among non-pharmacological methods in symptom control. As a result of studies conducted with different patient groups in the literature, it has been stated that acupressure reduces dyspnea and anxiety levels. In this study, five tools will be used: Patient Identification Form, Modified Borg Dyspnea Scale (MBS), Medical Research Council (MRC) Dyspnea Scale, Beck Anxiety Scale (BAÖ) and Patient Follow-up Schedule. Individuals will be applied acupressure once a day for two minutes at LI4, HT7, LU1, ST36 points, for a total of 20 sessions. It is of great importance for nurses to follow current care methods, include them in nursing care and improve themselves in this regard. No current study has been found in the literature investigating the effect of acupressure applied to individuals with COPD on dyspnea and anxiety. The purpose of this study is to determine the effect of acupressure applied to individuals with COPD on dyspnea and anxiety.

ELIGIBILITY:
Inclusion Criteria:

Patients who are literate,

Have moderate and severe stage COPD according to GOLD criteria,

Score 8 and above on the Beck Anxiety Inventory,

Patients who volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Patients using psychiatric medication (anxiolytic, antidepressant), Those with serious pulmonary, cardiological or malignant diseases, Those with vision and hearing problems, Those with communication problems, Those with nerve, soft tissue and vascular diseases in the areas where acupressure will be applied, Those with infections and surgical operations in the areas where acupressure will be applied, Patients in the exacerbation period were not included in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Effect of acupressure on dyspnea and anxiety in individuals with COPD | through study completion, an average of 1 year
  The Modified Borg Dyspnea Scale (MBS) was developed in 1982 by Gunnar Borg to define the intensity of physical activity. The original Borg scale is scored between 6-20. In 1986, the "American College of Sports Medicine" revised the scale by scoring between 0-10. Although the Modified Borg Scale is frequently used today to define the severity of exertional dyspnea, it is also a scale that can be used to evaluate the severity of resting dyspnea. The fact that there are various definitions in the Modified Borg Scale (MBS) makes it easier for patients to apply.
Effect of acupressure on dyspnea and anxiety in individuals with COPD | through study completion, an average of 1 year
  Medical Research Council Dyspnea Scale (MRC) The Medical Research Council (MRC) Dyspnea Scale was first used by Fletcher in 1952 to compare the severity of dyspnea during activity in people with and without lung disease. Later, the British Medical Research Council (MRC) introduced this scale in a more developed form to monitor the natural course of the disease. The dyspnea scale was created based on various physical activities that cause dyspnea. It consists of a total of 5 items and is a 1-5 point scale. The patient reads the scale options and selects the most appropriate degree that describes respiratory distress. In the MRC dyspnea scale, 1 describes the best dyspnea and 5 describes the worst. High scores on the scale indicate that the severity of shortness of breath is high.
Effect of acupressure on dyspnea and anxiety in individuals with COPD | through study completion, an average of 1 year
  Beck Anxiety Inventory The Beck Anxiety Inventory is a three-point Likert-type assessment scale consisting of 21 items that measures the frequency of anxiety symptoms experienced by an individual (0=none, 1=mild, 2=moderate, 3=severe). The highest score that can be obtained from the scale is 63. The high total score indicates the severity of anxiety. A score between 0-7 indicates "minimal anxiety", 8-15 indicates "mild anxiety", 16-25 indicates "moderate anxiety", and 26-63 indicates "severe anxiety". The scale was developed by Beck and his colleagues in 1988 and its validity and reliability in Turkish were performed by Ulusoy, Şahin, and Erkmen in 1996, and the Cronbach's α value was reported to be 0.93.
Effect of acupressure on dyspnea and anxiety in individuals with COPDThe schedule was prepared for the intervention group and will be used throughout the intervention. | through study completion, an average of 1 year
  Patient Follow-up Schedule Patients in the intervention group were followed up by phone calls every week to ensure regular and continuous acupressure application. The patient follow-up schedule was created by the researcher to record any problems with acupressure application and to provide the necessary information.
KOAH'lı bireylerde uygulanan akupresürün dispne ve anksiyete üzerine etkisi | through study completion, an average of 1 year
  The Modified Borg Dyspnea Scale (MBS) was developed in 1982 by Gunnar Borg to define the intensity of physical activity. The original Borg scale is scored between 6-20. In 1986, the "American College of Sports Medicine" revised the scale by scoring between 0-10. Although the Modified Borg Scale is frequently used today to define the severity of exertional dyspnea, it is also a scale that can be used to evaluate the severity of resting dyspnea. The fact that there are various definitions in the Modified Borg Scale (MBS) makes it easier for patients to apply.

CONTACTS AND LOCATIONS:
Overall Officials: songül k karadağ, Principal Investigator — çukurova universty
Locations (1):
- Cukurova University, Adana, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Pre- and post-implementation results of intervention and control group scales (statistical analysis). Participants' descriptive characteristics and participant consent form.
Supporting Information: ICF
Time Frame: Once published, the data is available indefinitely.
Access Criteria: data can be shared publicly.
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/